CLINICAL TRIAL: NCT03071861
Title: Mild Encephalopathy in the Newborn Treated With Darbepoetin (MEND)
Brief Title: Mild Encephalopathy in the Newborn Treated With Darbepoetin
Acronym: MEND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: University of Utah (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MEND 16-330
Record Dates: First submitted 2016-12-01; First posted 2017-03-07 (Actual); Results first posted 2023-07-25 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Neonatal Encephalopathy; Hypoxic-Ischemic Encephalopathy Mild
Keywords: darbepoetin; Brain Diseases
MeSH Terms: conditions — Brain Diseases | interventions — Darbepoetin alfa; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Darbepoetin Alpha (Experimental): IV,10 mcg/kg/dose, Darbepoetin Alpha, one dose at <24 hours of age
  Interventions: Drug: Darbepoetin Alfa
- Placebo (Placebo Comparator): IV, Normal saline (placebo dose), one dose at <24 hours of age
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Darbepoetin Alfa — Single dose of 10 mcg/kg Darbepoetin Alpha given IV at less than 24 hours of age
  Other Names: Darbe; Darbepoetin
  Arms: Darbepoetin Alpha
Drug: Normal Saline — Single dose of normal saline, IV, given at less than 24 hours of age
  Arms: Placebo

SUMMARY:
This is a Phase II multicenter placebo-controlled randomized, feasibility/safety trial. Infants >34 week gestational age with perinatal acidemia and mild neonatal encephalopathy on the modified Sarnat neurologic examination at less than six hours of age. Participants will be randomized to receive either one dose of Darbepoetin, or placebo within 24 hours of birth. Neurodevelopmental testing (Bayley (III or IV) and Gross Motor Function Assessment) will be performed at 24 months of age. Pharmacokinetics will be assessed on those infants that received Darbe.

DETAILED DESCRIPTION:
Therapeutic hypothermia (TH) is the standard of care for newborns diagnosed with moderate to severe neonatal encephalopathy (NE) presumably due to hypoxic ischemia. In order to be eligible for TH an infant must have perinatal acidemia and evidence of moderate or severe encephalopathy on a standardized neurologic examination (Sarnat). However, the majority of newborns with perinatal acidemia do not have a neurologic examination abnormal enough to be classified as moderate or severe NE. In a retrospective review, DuPont et al. found that as many as 20% of newborns with perinatal academia and mild NE have abnormal short-term outcomes such as seizures, death from progressive asphyxia insult, brain MRI findings consistent with NE, abnormal neurologic examination at discharge, gastrostomy tube feeding, or feeding difficulties. Preliminary data from a prospective trial investigating mild NE (PRIME study, NCT01747863) found that 39% had either abnormal electroencephalography at < 9h of age, an abnormal brain MRI finding, or abnormal neurological exam at discharge. Murray et al. recently reported on 5-year outcomes of infants with mild encephalopathy and showed that 25% had neurodevelopmental disability. These data suggest that mild NE likely carries a higher risk of impaired neurological outcome then reported previously. Thus it would appear that neuroprotective strategies would be beneficial in this group of infants. Preliminary data suggest that erythropoiesis stimulating agents (ESA) provide neuroprotection, and improve short and long-term neurologic outcome in neonatal brain injury. ESA may work through several mechanisms including reduced inflammation, limited oxidative stress, decreased apoptosis and white matter injury, as well as via pro-angiogenic and neurogenic properties. Darbepoetin alfa (Darbe), a recombinant human erythropoietin (EPO)-derived molecule has established safety and pharmacokinetics in newborns. Because Darbe has an extended circulating half-life with comparable biological activity to EPO, it has the advantage of requiring less frequent administration

ELIGIBILITY:
Inclusion Criteria: Infants will be eligible for the MEND trial if they have a gestational age > 34 weeks by best obstetric estimate, are <24 hours old and have evidence of mild encephalopathy as defined by Shankaran et al based on a modified Sarnat examination performed at <6 hours of age.

1. History of an acute perinatal event (abruption, cord prolapsed, severe fetal heart rate abnormality, or meconium staining)
2. Infant is evaluated for hypothermia therapy and DOES NOT meet clinical criteria for TH.
3. Infant has an IV for clinical treatment

Exclusion Criteria:

1. Moderate/Severe encephalopathy on modified Sarnat examination at < 6 hours of age
2. Major congenital and/or chromosomal abnormalities
3. Prenatal diagnosis of brain abnormality or hydrocephalus
4. Severe growth restriction (< 3%)
5. Central venous hematocrit >65%, platelet count >600,000/dL, and/or neutropenia (ANC<500 μL)
6. ECMO
7. Infant judged critically ill and unlikely to benefit from neonatal intensive care by the attending neonatologist

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2022-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara L DuPont, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Darbepoetin Alpha | Placebo
Started | 13 | 15
Completed | 12 | 14
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: 13 infants were enrolled in the Darbe arm and 15 were enrolled in the placebo arm
Groups:
- Total: Total of all reporting groups
Arm/Group | Darbepoetin Alpha | Placebo | Total
Number analyzed (Participants) | 13 | 15 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 13 | 15 | 28
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 39 (1.9) | 39 (1.5) | 39 (1.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 7 | 13
  Male | 7 | 8 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 13 | 15 | 28
gestational age less than 36 weeks [Count of Participants; unit: Participants] | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Normal Neurodevelopment
Description: The Bayley III and Neuromuscular Assessment were completed between 9-12 months of age. Subjects were abnormal if they had a Bayley III score of less than 70 and/or an abnormal neurological examination.
Time Frame: 9 - 12 months of age
Population: one infant was lost to follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alpha | Placebo
Number analyzed (Participants) | 13 | 14
Participants | 13 | 14

2. Secondary Outcome: Percent of Infants With Adverse Events
Description: Potential adverse events such as (but not limited to) alterations in blood pressure, secondary infections, neutropenia, thrombotic/vascular events, hematologic events (platelets, Hct level, polycythemia), and hepatic/renal function that are outside of normal range for the study population.
Time Frame: 30 days or until hospital discharge whichever comes first
Population: There were NO adverse events reported
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alpha | Placebo
Number analyzed (Participants) | 13 | 15
Participants | 0 | 0

3. Secondary Outcome: Percent of Infants With Seizures
Description: development of clinical or electrographic seizures
Time Frame: 30 days or until hospital discharge whichever comes first
Population: Patients with seizures after study enrolment
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alpha | Placebo
Number analyzed (Participants) | 13 | 15
Participants | 0 | 0

4. Secondary Outcome: Percentage of Infants Who Need Gavage Feeds or Gastrostomy at Discharge Home
Description: Infants who require tube feedings at discharge
Time Frame: 30 days or until hospital discharge whichever comes first
Population: Discharge feeding method
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alpha | Placebo
Number analyzed (Participants) | 13 | 15
Participants | 0 | 0

5. Other Pre Specified Outcome: Percent With Seizures
Description: development of clinical or electrographic seizures
Time Frame: 24 months of age
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Percent With Failure to Thrive
Description: Growth at <3%
Time Frame: 9 months of age
Population: 27 infants were followed at 9 months of age. One infant in the placebo arm was lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alpha | Placebo
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

7. Other Pre Specified Outcome: Percent With Hearing Impairment
Description: Child requires a hearing device
Time Frame: 9 months of age
Population: one infant was lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alpha | Placebo
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

8. Other Pre Specified Outcome: Percent With Vision Impairment
Description: requires corrective lenses
Time Frame: 9 months of age
Population: one infant was lost to follow up
Measure: Count of Participants; unit: Participants
Arm/Group | Darbepoetin Alpha | Placebo
Number analyzed (Participants) | 13 | 14
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: birth to 9 months
Description: No subject died during this trial.
Arm/Group | Darbepoetin Alpha | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 0/13 | 0/15

LIMITATIONS AND CAVEATS:
pK analysis has not been completed yet.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-18): https://cdn.clinicaltrials.gov/large-docs/61/NCT03071861/Prot_SAP_007.pdf
  • Informed Consent Form (2018-12-04): https://cdn.clinicaltrials.gov/large-docs/61/NCT03071861/ICF_008.pdf